CLINICAL TRIAL: NCT03685513
Title: One Year Clinical Evaluation of Milled BioHPP Polyetheretherketone (PEEK)-Based Versus Metal Ceramic Single Crowns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdelrahman Soliman Elsayed Badran, Resident, Fixed Prosthodontics Department, Faculty of Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-09-30
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Single Posterior Crowns; Badly Decayed Teeth, Teeth Restored With Large Filling Restorations or Endodontically Treated Teeth; Malformed Teeth, Malposed Teeth (Tilted, Over-erupted, Rotated, Etc.) or Spacing Between Posterior Teeth
MeSH Terms: conditions — Tooth, Nonvital; Tooth Abnormalities | interventions — Melanocyte-Stimulating Hormones

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metal ceramic single posterior crowns (Active Comparator): Metal copings veneered with feldspathic porcelain
  Interventions: Other: Metal ceramic single posterior crowns
- BioHPP PEEK-based single posterior crowns (Experimental): BioHPP PEEK copings veneered with composite resin
  Interventions: Other: BioHPP PEEK-based single posterior crowns

INTERVENTIONS:
Other: BioHPP PEEK-based single posterior crowns — BioHPP PEEK is 20% ceramic reinforced, semicrystalline, thermoplastic and radiolucent polymer for extreme durability especially for frameworks for fixed and removable dental prostheses. It has many advantages as low density, light weight, shock absorber, biocompatible and venerable with composite resin.
  Arms: BioHPP PEEK-based single posterior crowns
Other: Metal ceramic single posterior crowns — Standard metal coping veneered with glass ceramics
  Other Names: Porcelain fused to metal (PFM) or Ceramo-metallic
  Arms: Metal ceramic single posterior crowns

SUMMARY:
Although the metal-ceramic system is still widely used to fabricate crowns and fixed partial dentures and is considered as the standard treatment in dentistry, aesthetic concerns have stimulated the development of new dental tooth-colored systems as PEEK.

BioHPP PEEK is 20% ceramic reinforced, semicrystalline, thermoplastic and radiolucent polymer for extreme durability especially for frameworks for fixed and removable dental prostheses. It has many advantages as low density, light weight, shock absorber, biocompatible and venerable with composite resin.

The aim of this study is to evaluate the clinical performance of milled BioHPP PEEK-based single crowns and compare them to metal-based single crowns.

ELIGIBILITY:
Inclusion Criteria:

1. From 18-50 years old, be able to read and sign the informed consent document.
2. Have no active periodontal or pulpal diseases, have teeth with good restorations
3. Psychologically and physically able to withstand conventional dental procedures
4. Patients with teeth problems indicated for single posterior crowns:

   1. Badly decayed teeth
   2. Teeth restored with large filling restorations
   3. Endodontically treated teeth
   4. Malformed teeth
   5. Malposed teeth (Tilted, over-erupted, rotated, etc.)
   6. Spacing between posterior teeth
5. Able to return for follow-up examinations and evaluation

Exclusion Criteria:

1. Patient less than 18 or more than 50 years
2. Patient with active resistant periodontal diseases
3. Patients with poor oral hygiene and uncooperative patients
4. Pregnant women
5. Patients in the growth stage with partially erupted teeth
6. Psychiatric problems or unrealistic expectations
7. Lack of opposing dentition in the area of interest

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Fracture | 1 year
  Measured using modified USPHS criteria

SECONDARY OUTCOMES:
Marginal adaptation | 1 year
  Measured using modified USPHS criteria

OTHER OUTCOMES:
Patient Satisfaction | 1 year
  Measured using modified USPHS criteria

IPD SHARING:
Plan to Share IPD: Undecided